CLINICAL TRIAL: NCT04566705
Title: Uterine Rupture During Labor Among Women With a Prior Cesarean Delivery : Risks Factors, Maternal and Perinatal Outcomes
Brief Title: Uterine Rupture During Labor Among Women With a Prior Cesarean Delivery
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL20_0142
Record Dates: First submitted 2020-09-14; First posted 2020-09-28 (Actual); Last update posted 2020-11-18 (Actual); Status verified 2020-09

CONDITIONS: Uterine Rupture; Mode of Delivery
Keywords: Risks factors; Uterine rupture after a previous cesarean delivery; Vaginal birth after cesarean; Prior cesarean; Perinatal outcome
MeSH Terms: conditions — Uterine Rupture

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Women with uterine rupture: Women with uterine rupture
- Women without uterine rupture: Women without uterine rupture
  Interventions: Other: Risks factors, maternal and neonatal outcomes/complications

INTERVENTIONS:
Other: Risks factors, maternal and neonatal outcomes/complications — Risks factors, maternal and neonatal outcomes/complications
  Groups: Women without uterine rupture

SUMMARY:
Although a rare event, uterine rupture during labour is one of the most serious obstetric complications because of the dramatic maternal-fetal consequences that can result.

Identifying the risk factors associated with uterine rupture would enable gynecologists to provide patients with risks of uterine rupture in the event of attempted vaginal delivery.

The aim of our study is to determine risks factors for uterine rupture during labour in patients with a previous cesarean delivery who have not given birth since and to assess the occurrence of maternal-fetal comply-cations compared to patients with a previous cesarean delivery without uterine rupture.

ELIGIBILITY:
Inclusion criteria:

* Singleton pregnancy > 24 weeks of gestation
* Second or multiparous with a previous cesarean section without vaginal delivery since
* Cephalic presentation or completed breech
* Uterine rupture during labor

Exclusion criteria:

* Incomplete uterine rupture
* Multiple gestation
* Transverse presentation or complete breech
* Vaginal delivery after cesarean
* Non-low transverse cesarean section
* Placenta praevia
* Antepartum intrauterine fetal death
* History of uterine surgery (myomectomy)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women with uterine rupture after previous cesarean delivery versus women without uterine rupture after previous cesarean delivery
Sampling Method: Non-Probability Sample
Enrollment: 95 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-04-01 (Actual)

PRIMARY OUTCOMES:
Assess the risks factors of uterine rupture | 1 day
  Assess the risks factors of uterine rupture
  Assess the risks factors of uterine rupture using obstetric measures

SECONDARY OUTCOMES:
Number of Participants with Assess the maternal and perinatal complications and outcomes | 1 day
  Number of Participants withAssess the maternal and perinatal complications and outcomes : looking for maternal complications (chorioamnionitis , transfusion, post-partum hemorrhage, surgery for blad-der wound, maternal death,…) and neonatal comply-cations (apgar<7 at 5minutes, pH <7,15, neonatal intein-sive care unit and perinatal death)

CONTACTS AND LOCATIONS:
Overall Officials: Florent FUCHS, PUPH, Study Director — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC